CLINICAL TRIAL: NCT00299611
Title: A Double-Blind Augmentation Study of LEvetiracetam in Obsessive Compulsive Disorder
Brief Title: Augmentation Study of Levetiracetam in Obsessive Compulsive Disorder
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decided to terminate the study due to budget consideration
Sponsor: Duke University (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Wei Zhang/ Director of Anxiety and Traumatic Stress Program, DUMC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00008596
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2010-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Anxiety; Pharmacotherapy; Sertraline; Levetiracetam
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders | interventions — Sertraline; Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Levetiracetam
  Interventions: Drug: Sertraline; Drug: Levetiracetam
- 2 (Placebo Comparator): there is no active ingredient in the pills.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline — Tablets, 50mg each, (1-3TABLETS/DAY) during the Open-label phase for first 8 wks.
  Other Names: Zoloft
  Arms: 1
Drug: Levetiracetam — Tablets, dosage 500mg each tablet (1-4tablets/day)for 8 wks during the 2nd phase of the study.
  Other Names: Keppra
  Arms: 1
Drug: Placebo — Tablets, No active ingredient, (1-4tablets/day) for 8 wks during the 2nd phase of the study.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Levetiracetam augmentation relative to Placebo in SSRI non-remitters with obsessive compulsive disorder. The hypothesis is that anxiolytic effect of Levetiracetam is more beneficial when adding with a SSRI.

DETAILED DESCRIPTION:
This is an investigator-initiated, single-site study, consisting of two phases: 8 weeks of open-label treatment with sertraline (50mg-150mg/day) in patients iwth OCD.At week 8, those who have failed to achieve remission will be continued on sertraline and will be randomized to receive Levetiracetam (500mg-2000mg/day) or Placebo for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-65
* primary diagnosis of OCD based on DSM-IV criteria and assessed by the MINI International Neuropsychiatric Interview
* Yale-Brown Obsessive-Compulsive Scale (YBOCS) score of at least 16 or greater on screening
* Ability to provide written consent form

Exclusion Criteria:

* Any primary DSM-IV Axis I disorder other than OCD
* Substance abuse during the last 6 months
* A clinically unstable medical condition or clinically significant laboratory abnormalities
* Suicidal risk or serious suicidal attept during the last year
* Concurrent use of psychotropic medication including benzodiazepines, barbituates, antiepileptic drugs, antidepressants, buspirone, dietary supplements or herbal or homeopathic remedies with psychotropic effects
* Recent (within the last 3 months) initiation of cognitive behavioral therapy
* Failure of previous trial of levetiracetam at 2000 mg/day
* Pregnancy or lactation
* Women of childbearing potential who are unwilling to practice an acceptable method of contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-improvement (CGI-I) | 24 wks

SECONDARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (YBOCS) | 24 wks
Hospital Anxiety and Depression Scale | 24 wks
Sheehan Disability Scale (SDS) | 24 wks

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Ellingrod VL. Pharmacotherapy of primary obsessive-compulsive disorder: review of the literature. Pharmacotherapy. 1998 Sep-Oct;18(5):936-60. PMID 9758307
- [Background] Sasson Y, Zohar J, Chopra M, Lustig M, Iancu I, Hendler T. Epidemiology of obsessive-compulsive disorder: a world view. J Clin Psychiatry. 1997;58 Suppl 12:7-10. PMID 9393390
- [Background] Steketee G. Disability and family burden in obsessive-compulsive disorder. Can J Psychiatry. 1997 Nov;42(9):919-28. doi: 10.1177/070674379704200902. PMID 9429061
- See also: Related Info — http://dukehealth.org
- See also: Related Info — http://clinicaltrials.gov
- See also: Related Info — http://psychiatry.mc.duke.edu/Research/Research.html